CLINICAL TRIAL: NCT04937673
Title: Camrelizumab Combined With Chemotherapy for Neoadjuvant Treatment of Locally Advanced Thoracic Esophageal Squamous Cell Carcinoma：A Phase II Clinical Study to Explore the Relationship Between Biomarkers and Efficacy
Brief Title: The Neoadjuvant Treatment of Locally Advanced Thoracic Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Director, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-EC-II-005
Record Dates: First submitted 2021-05-28; First posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Thoracic Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camrelizumab+ Paclitaxel+ Cisplatin (Experimental): The subjects were randomly divided into the group of camrelizumab combined with paclitaxel and cisplatin or the group of camrelizumab combined with albumin bound paclitaxel and cisplatin according to the ratio of 1:1. Esophageal cancer resection was performed after 3 cycles of medication (the researchers decided the follow-up treatment according to the postoperative pathological situation). At the end of the treatment, the patients were followed up for safety and effectiveness.
  Interventions: Drug: Camrelizumab+ Paclitaxel+ Cisplatin
- Camrelizumab+ Albumin bound paclitaxel+ Cisplatin (Experimental): The subjects were randomly divided into the group of camrelizumab combined with paclitaxel and cisplatin or the group of camrelizumab combined with albumin bound paclitaxel and cisplatin according to the ratio of 1:1. Esophageal cancer resection was performed after 3 cycles of medication (the researchers decided the follow-up treatment according to the postoperative pathological situation). At the end of the treatment, the patients were followed up for safety and effectiveness.
  Interventions: Drug: Camrelizumab+Albumin bound paclitaxel+Cisplatin

INTERVENTIONS:
Drug: Camrelizumab+Albumin bound paclitaxel+Cisplatin — Camrelizumab: intravenous drip, fixed dose 200 mg, D1, repeated once every 3 weeks.
  Albumin bound paclitaxel: 130 mg / m2, intravenous drip for 30 minutes, D1, D8, repeated every 3 weeks.
  Cisplatin: 75 mg / m2, intravenous drip for 120 minutes, D1, repeated every 3 weeks.
  Arms: Camrelizumab+ Albumin bound paclitaxel+ Cisplatin
Drug: Camrelizumab+ Paclitaxel+ Cisplatin — Camrelizumab: intravenous drip, fixed dose 200 mg, D1, repeated once every 3 weeks.
  Paclitaxel: 80 mg / m2, intravenous drip for 180 minutes, D1, D8, repeated every 3 weeks.
  Cisplatin: 75 mg / m2, intravenous drip for 120 minutes, D1, repeated every 3 weeks.
  Arms: Camrelizumab+ Paclitaxel+ Cisplatin

SUMMARY:
This is a randomized, open, two arm phase II clinical study. 40 patients are included in the exploratory study. The dominant population with higher biomarker positive / IO score was identified to provide the basis for the later phase III study. The subjects were randomly divided into the group of camrelizumab combined with paclitaxel and cisplatin or the group of camrelizumab combined with albumin bound paclitaxel and cisplatin according to the ratio of 1:1. The treatment cycle was every 3 weeks. The curative effect was evaluated when the treatment cycle was 2, and the resection of esophageal cancer was considered after 3 cycles. Postoperative adjuvant therapy was based on the patient's condition and surgical results; For patients with R0 resection, postoperative adjuvant treatment is not recommended. For patients with R1 / R2 resection, multi-disciplinary joint discussion and consultation are recommended to propose individualized comprehensive treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years old, male or female;
2. Esophageal squamous cell carcinoma was confirmed by pathology (except for cervical and Suprathoracic tumors that could not be operated);
3. Patients with resectable esophageal squamous cell carcinoma with clinical stage T3-T4a or TxN + M0 (except T4b);
4. ECOG PS score was 0-1;
5. There was at least one measurable lesion (according to recist1.1) or unmeasurable lesion that could be evaluated, and the imaging diagnosis time was ≤ 21 days;
6. The expected survival time was more than 3 months;
7. The function of the main organs was normal, and there were no serious blood, heart, lung, liver, kidney, bone marrow and other functional abnormalities and immunodeficiency diseases. The laboratory examination meets the following requirements:

   1. Hemoglobin (Hb) ≥ 90g / L;
   2. WBC ≥ 3.0 × 109/L； Neutrophil count (NEUT) ≥ 1.5 × 109/L；
   3. Platelet count (PLT) ≥ 100 × 109/L；
   4. Serum creatinine (SCr) ≤ 1.5 times the upper limit of normal (ULN) or creatinine clearance rate ≥ 50 ml / min (Cockcroft Gault formula);
   5. Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN);
   6. The levels of AST and ALT were less than 2.5 times the upper limit of normal (ULN);
8. There was no active bleeding or thrombosis

   1. International normalized ratio INR ≤ 1.5 × ULN；
   2. Partial thromboplastin time APTT ≤ 1.5 × ULN；
   3. Prothrombin time Pt ≤ 1.5ULN;
9. The patients with normal or mild to moderate abnormal lung function (VC% > 60%, FEV1 > 1.2L, FEV1% > 40%, DLco> 40%) could tolerate esophagectomy;
10. The fertile female subjects were required to conduct blood pregnancy test within 72 hours before the first administration, and the result was negative, and voluntarily used appropriate contraceptive methods during the observation period and within 90 days after the last administration of the study drug; For men, surgical sterilization or consent to appropriate contraceptive methods during the observation period and within 90 days after the last administration of the study drug should be used.
11. The subjects voluntarily joined the study and signed the informed consent form (ICF);
12. The patients with good compliance were expected to follow up the efficacy and adverse events / reactions according to the protocol requirements.

Exclusion Criteria:

1. Subjects who have received or are receiving additional chemotherapy, radiotherapy, targeted or immunotherapy;
2. Any active autoimmune disease or history of autoimmune disease (such as interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (can be included after hormone replacement therapy)); The subjects with childhood asthma who had been completely relieved and did not need any intervention or vitiligo in adulthood could be included, but the subjects who needed bronchodilator for medical intervention could not be included;
3. Patients with congenital or acquired immune deficiency, such as human immunodeficiency virus (HIV) infection, active hepatitis B (HBV DNA ≥ 500 IU / ml), hepatitis C (HCV antibody positive and HCV-RNA higher than the detection limit of the analytical method), or co infection of hepatitis B and hepatitis C;
4. Immunosuppressive drugs were used within 14 days before the first use of the study drug, excluding nasal and inhaled corticosteroids or physiological doses of systemic corticosteroids;
5. Live attenuated vaccine was inoculated within 4 weeks before the first administration or during the study period;
6. Patients with hypertension who can not be reduced to normal range after antihypertensive drug treatment (systolic blood pressure ≤ 140 mmHg / diastolic blood pressure ≤ 90 mmHg);
7. Subjects with uncontrollable clinical cardiac symptoms or diseases, such as (1) heart failure of NYHA II or above (2) unstable angina pectoris (3) myocardial infarction within 1 year (4) clinically significant supraventricular or ventricular arrhythmia requiring clinical intervention;
8. Severe infection (e.g. need for intravenous antibiotics, antifungal or antiviral drugs) occurred within 4 weeks before the first administration, or fever of unknown origin > 38.5% occurred during the screening period / before the first administration；
9. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation is known;
10. Pregnant or lactating women; The fertile subjects were unwilling or unable to take effective contraceptive measures;
11. Other malignant tumors were found in the past or at the same time, but the cured basal cell carcinoma of skin, carcinoma in situ of cervix and carcinoma in situ of breast were excluded;
12. Known to have allergic history to the drug components of this protocol;
13. Other situations considered unsuitable by the researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
biomarkers related to pCR | 9 weeks
  t has a good value in predicting the efficacy of immunotherapy, and is helpful for the accurate formulation of treatment plan and the accurate evaluation of prognosis of patients with esophageal cancer.

SECONDARY OUTCOMES:
Objective Response Rate | 9 weeks
  Assess ORR, defined as Investigator-assessed CR + PR, per RECIST 1.1.
Disease Control Rate | 9 weeks
  Percentage of patients with CR/PR/SD in the number of patients that whose tumour can be evaluated.
Disease free survival | Time from randomization to patient's tumor progression or death
  The DFS will be defined as the time of patients alive without local recurrence or distant metastasis of disease from the date of the administration of treatment.
Overall Survival | The time from the beginning of randomization to death due to any cause.
  OS is defined as the time from registration to death due to any cause, or censored at date last known alive. Measured by the method of Kaplan and Meier
Safety | from first treatment to 90 days after esophagectomy
  Adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Department of GI Oncology, Peking University Cancer Hospital,, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No